CLINICAL TRIAL: NCT04250233
Title: Prospective Observational Study of Postoperative Respiratory Rate After Cesarean Delivery Among a Convenience Sample of Women Undergoing Spinal Anesthesia With and Without Neuraxial Opioids
Brief Title: Respiratory Rate After Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: TASMC-2020-CFW-608-19-CTIL
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cesarean Delivery; Neuraxial Opioids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard neuraxial opioids: Standard neuraxial anesthesia for cesarean delivery (heavy bupivacaine 10 mg; fentanyl 10-25 mic; and low dose intrathecal morphine
  Interventions: Device: Respiratory Monitor
- Non standard neuraxial opioids: Non standard low-dose morphine group (with heavy bupivacaine 10 mg; fentanyl 10-25 mic)
  Women are offered - if they prefer not to receive low dose morphine, the option of either ultra-low dose morphine or no morphine - instead they can receive postoperative bilateral quadratus lumborum block (QLB), TAP or erector spinus block.
  Interventions: Device: Respiratory Monitor

INTERVENTIONS:
Device: Respiratory Monitor — All women receive a respiratory rate monitor after cesarean delivery. We anticipate that at least 30 women will receive standard dose neuraxial block, and aim to have a cohort of 20-30 women who receive non-standard dose (Group 20 in order to compare respiratory rates.

SUMMARY:
The study proposal summarizes aspects related to respiratory rate in women who undergo spinal anesthesia for cesarean delivery who receive or do not receive neuraxial opioids

DETAILED DESCRIPTION:
Respiratory monitoring device will be used to count respiratory rate continuously, as opposed to the intermittent nursing respiratory rate (RR) counts once per hour. The device counts respiration (RR) using a sticker placed by on the neck to detect vibrations made by respiration. This overcomes the specific limitation of capnography that requires wearing the nasal cannula.

Prospective, observational study with institutional review board (IRB) approval. Women who undergo elective cesarean delivery under neuraxial block receive neuraxial opioids for postoperative analgesia.

Potential study recruits will be approached prior to the cesarean delivery anesthesia assessment. Suitable women will be informed that neuraxial morphine is the gold-standard analgesia, however many women suffer nausea, vomiting and pruritus (itching) and may prefer an alternative analgesic or a lower dose of morphine. All women will receive intrathecal fentanyl as an adjuvant to the bupivacaine anesthesia. This fentanyl may also cause pruritus however this is limited to the 2-hour duration of the effect of the fentanyl.

Women will be offered standard neuraxial anesthesia for cesarean delivery (heavy bupivacaine 10 mg; fentanyl 10-25mic; and low dose intrathecal morphine mic). Alternatively, women will be offered an alternative anesthesia option: 1) heavy bupivacaine 10 mg; fentanyl 10-15 mic with an ultra-low dose, 50 mic of morphine, or 2) heavy bupivacaine 10 mg; fentanyl 10-25 mic without intrathecal morphine + postoperative bilateral quadratus lumborum block (QLB), transversus abdominis plane (TAP) or erector spinus block (ESP). For patients who select block without intrathecal morphine, the choice of block will depend on anesthesiologist's decision.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class II or III
* age between 18 and 50
* gestational age greater than 37 completed weeks
* singleton pregnancy. In contrast to previous studies
* we do not plan to exclude obese women and those with suspected sleep apnea.

Exclusion Criteria:

* Contraindication for epidural analgesia (bleeding diathesis, neuropathy, severe scoliosis, previous spine surgery, local anesthetic allergy)
* narcotic administration in the previous 2 hours
* inability to adequately understand the consent form
* moderate-severe asthma, inability to receive morphine
* sensitivity to sticker
* skin conditions.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female pregnant
Study Population: Women undergoing elective cesarean delivery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Respiratory rate ≤8 | up to 24 hours
  Our primary study aim is to report the number of women with RR≤8 at any time point after the cesarean delivery using the continuous respiratory monitoring device.

SECONDARY OUTCOMES:
respiratory rate per min | up to 24 hours
  To report the minimum/maximum values for: respiratory rate per min among women who receive standard low dose neuraxial opioids for postoperative analgesia and to compare to other groups
oxygen saturation | up to 24 hours
  - To report the minimum/maximum values for: oxygen saturation for women who undergo cesarean delivery and receive standard low-dose neuraxial opioids and to compare to other groups.
heart rate | up to 24 hours
  - To report the minimum/maximum values for: heart rate for women who undergo cesarean delivery and receive standard low-dose neuraxial opioids and to compare to other groups.
apnea | up to 24 hours
  - To report the frequency of apnea for women who undergo cesarean delivery and receive standard low-dose neuraxial opioids and to compare to other groups.
side effects | up to 24 hours
  incidence ie no of women with and without pruritus, nausea, vomiting, other side effects of analgesia and compare between groups
additional analgesia | up to 24 hours
  post operative analgesia used for each patient in 24 hours (paracetamol, ibuprofen, optalgin, other) and compare between groups
antiemetic | up to 24 hours
  antiemetic administration for each patient in 24 hours and compare between groups - women with and without resp depression
duration of monitor period | up to 24 hours
  duration of use of monitor (pulse oximeter, RR, HR) - all and each of the components
nurse outcomes | up to 24 hours
  nurse measured outcomes - the number of the RR recorded, and compare between groups - women with and without resp depression
patient experience | up to 24 hours
  patient will be asked for verbal descriptions after being prompted - how did you find the experience of using the device to assess patient experience of the device (discomfort, nursing interference, mobility interference, family visit interference, itchy, nausea, others)
patient anesthesia selection | up to 24 hours
  To report the number of women who select each of the anesthesia modalities offered (standard low dose; ultra-low dose morphine; or truncal nerve block (QLB/TAP/ESP).

CONTACTS AND LOCATIONS:
Locations (1):
- Tel AViv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No